CLINICAL TRIAL: NCT05772858
Title: Family Therapy Training and Implementation Platform (FTTIP): An Innovative Web-based Tool for Long-term Practice Improvement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Training and Implementation Associates (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1R43MH115547-01A1 (NIH)
Record Dates: First submitted 2023-02-23; First posted 2023-03-16 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Traditional Face to Face Training; Family Therapy Training and Implementation Platform (FTTIP)
Keywords: Mental health; Family therapy; Mental health training
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: 150 therapists will be randomly assigned to be trained by either the Family Therapy Training and Implementation Platform (FTTIP) or a Traditional in person Training as Usual (TAU). 150 families will all receive the Culturally Informed Flexible and Family based Treatment for Adolescents. 30 agency leaders will be randomly assigned to Family Therapy Training and Implementation Platform (FTTIP) agency readiness consultation or Agency readiness consultation as usual.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Family Therapy Training and Implementation Platform (FTTIP) (Experimental): Participants will be trained for 20 hours on an online platform practicing family therapy competencies with animated families and provided recorded video responses to receive feedback from trainers.
  Interventions: Other: Training on CIFFTA competencies using Family Therapy Training and Implementation Platform (FTTIP)
- Traditional in person Training as Usual (Active Comparator): Participants will attend 20 hours of a traditional in person training learning about the family therapy evidenced based treatment.
  Interventions: Other: Training on CIFFTA competencies using Training and Coaching as Usual (TCAU).
- Culturally Informed and Flexible Family-Based Treatment for Adolescents (CIFFTA). (Experimental): All of the 150 families will receive Family Therapy, Individual Therapy, and Psycho-educational Modules, delivered over 16 weeks in a two session (60 minutes each) per week format.
  Interventions: Other: Culturally Informed and Flexible Family-Based Treatment for Adolescents (CIFFTA).
- Agency Readiness Consultation- Family Therapy Training and Implementation Platform (FTTIP) (Experimental): Agency leaders assigned to this condition will complete an online assessment of agency readiness, participate in a webinar and live discussion, complete an online meeting with leaders and clinical supervisors
  Interventions: Other: Agency Readiness Consultation- Family Therapy Training and Implementation Platform (FTTIP)
- Agency Engagement and Orientation as Usual (Active Comparator): Agency leaders assigned to this condition will receive a traditional engagement of leadership at their agency including a description of study procedures and engagement with study team.
  Interventions: Other: Agency Engagement and Orientation as Usual

INTERVENTIONS:
Other: Training on CIFFTA competencies using Family Therapy Training and Implementation Platform (FTTIP) — An Innovative Web-based Tool to train mental health therapists in family therapy competencies with animated families and provided recorded video responses to receive feedback from trainers.
  Arms: Family Therapy Training and Implementation Platform (FTTIP)
Other: Training on CIFFTA competencies using Training and Coaching as Usual (TCAU). — Therapists receive training using the traditional face to-face training method for 2.5 days followed by coaching.
  Arms: Traditional in person Training as Usual
Other: Culturally Informed and Flexible Family-Based Treatment for Adolescents (CIFFTA). — CIFFTA has three major components: Family Therapy, Individual Therapy, and Psycho-educational Modules, delivered over 16 weeks in a two session (60 minutes each) per week format. One session will typically be a family session which may include Family Therapy or Psychoeducational modules designed for the family or parents alone. The other session is typically with the adolescent alone which may include individual treatment or Psycho-educational modules designed for the adolescent.
  Arms: Culturally Informed and Flexible Family-Based Treatment for Adolescents (CIFFTA).
Other: Agency Readiness Consultation- Family Therapy Training and Implementation Platform (FTTIP) — The FTTIP agency readiness work begins with a pre-recorded FTTIP introduction webinar presented separately to each agency which presents overall goals of the project and the different FTTIP components, and key decisions agencies often make when seeking to sustain a new EBT.
  Arms: Agency Readiness Consultation- Family Therapy Training and Implementation Platform (FTTIP)
Other: Agency Engagement and Orientation as Usual — Work with the agency leaders will consist of the traditional engagement of the leadership so that they agree to collaboration with the study team, with the training team, and with the study procedures.
  Arms: Agency Engagement and Orientation as Usual

SUMMARY:
The goal of this clinical trial is to compare whether mental health therapists trained by a Family Therapy Training and Implementation Platform (FTTIP) or those trained in traditional face-to-face training differ on learning key family therapy domains, including competencies, agency readiness, and client outcomes. The main questions it aims to answer are:

* Will 75 FTTIP mental health therapists show improvement in all core family therapy competencies that are not inferior to 75 providers receiving traditional in person family therapy training?
* Will 150 families (child, parent, dyad) receiving CIFFTA family therapy show adequate retention in treatment therapeutic alliance and significant pre-post treatment improvements on family environment and presenting problems?
* Will 15 agency leaders receiving FTTIP agency readiness consultations show more pre and post change in agency readiness and knowledge than 15 leaders receiving agency engagement as usual?

Participants will participate in:

* Complete pre and post surveys
* 20 hours of training in an evidenced based family therapy treatment
* 24 weeks of biweekly coaching to implement the treatment
* 24 weeks of implementation of the treatment with one family
* Agency leaders will complete 2 weeks of organizational readiness engagement

Researchers will compare the Family Therapy Training and Implementation Platform (FTTIP) and traditional face-to-face training to see if FTTIP is not inferior to traditional training in key domains, including competencies, agency readiness, and client outcomes in mental health therapists.

DETAILED DESCRIPTION:
Family therapy has emerged as one of the most efficacious interventions for child and adolescent behavioral and psychiatric issues and for chronic health conditions. However, widespread implementation of family therapy is often hampered by high training costs, re-training needs following staff turnover, low agency readiness to support new practices, and training strategies that lack ongoing implementation support and are prohibitively expensive. To better address the treatment needs of children and families, and to address long standing training and implementation challenges, we developed an innovative Family Therapy Training and Implementation Platform (FTTIP). FTTIP: 1) is guided by advances in implementation science, agency readiness, and knowledge of what it takes to sustain an evidence-based treatment; 2) uses adaptive training and consultation processes that provide a dynamic and data-driven procedure in which a competency is taught, measured, and the success or failure of the learning informs the next step of training in real time; 3) provides interactive practice of skills in which the trainee records interventions in response to simulation and receives personalized feedback; and 4) provides optional learning paths that allow the learner to explore additional ways to master the skills. Our Phase I study demonstrated the feasibility of FTTIP and set the stage for a fully-powered multisite Phase II Randomized Controlled Trial that will investigate whether FTTIP is "not inferior" to traditional face-to-face training on all key domains, including trainee competencies, agency readiness, and client outcomes. The Phase II study aims to: 1) Complete learning, practice and competency testing paths that provide the learner multiple learning options and to increase the dynamic nature of the platform; 2) Demonstrate that 75 FTTIP trainees show improvement in all core family therapy competencies that are not inferior to 75 providers receiving traditional in-person family therapy training as tested using pre and post training measures in a clinical trial; 3) Demonstrate that 150 families (child/parent dyad) receiving CIFFTA family therapy show adequate retention in treatment, therapeutic alliance, and significant pre-post treatment improvements on family environment and presenting problems; 4) Establish the process (e.g., initiation and delays in training new staff) and cost associated with training in each of the two conditions; 5) Demonstrate that 15 agency leaders receiving FTTIP agency readiness consultations show more pre and post change in agency readiness and knowledge than 15 leaders receiving agency engagement as usual. FTTIP's commercial application is that national, state, and local treatment services funders and providers will find FTTIP to be a highly cost effective, flexible, and engaging way to improve the quality of their evidence-based treatments (EBTs). By better preparing the nation's workforce on EBTs, and providing the support and coaching they need to reach full mastery, our FTTIP product has the potential to significantly improve the wellbeing and mental health in our nation and internationally.

ELIGIBILITY:
Inclusion Criteria:

* 150 Bachelor's level counselors with 2 years of experience or Master's level counselors and therapists who have not had family therapy training in the past year and who are broadly representative of the potential trainees in the general population, including educational background and job experience with different client populations (e.g., varied demographics and presenting problems). All therapists must be actively providing treatment to youth and be willing to deliver the family intervention to at least one family during the project period.
* For each trainee that is part of the research study, we will select one client family (1 child and 1 caregiver) that we will assess and follow during the study. Once a trainee completes training and begins coaching, the next child/family that is assigned to the trainee, meets criteria for CIFFTA, and consent/assents to participate will be considered a participant in the study. The child must be between the ages of 11-18 years. Other than that, there are no exclusion of any specific age or age range group in the rest of the study participants (agency leaders, counselors)
* 30 leaders will be randomized to the two conditions. To be included in the study, agency leaders must have the authority to allocate agency resources (e.g., giving trainees protected time to participate in training activities, allowing smaller caseloads as they begin implementation) and be willing to participate in agency readiness and implementation consultation.

Exclusion Criteria:

* We are not limiting inclusion of any group by sex/gender, race, and/or ethnicity
* Agencies that are unwilling to participate in all study activities, that have nontraditional funding sources (e.g., totally charity funded), or that are so small they cannot assign sufficient counselors to the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Retention in family therapy as measured by the number of sessions received by each study family | Post therapy at 24 weeks
  A critically important measure when working with underserved populations are indicators of staying in treatment (avoiding premature termination). The Retention measure will document the number of sessions received by each study family.
Change from pre therapy to post therapy treatment in family cohesion and family conflict as measured by the Family Environment Scale | Pre therapy (at baseline) and post therapy at 24 weeks
  This study will utilize two subscale of the Family Environment Scale, Family Cohesion and Family Conflict. Each subscale consists of 9 true-false items yielding scores from 0-9. The scales have been very useful in family therapy research and has strong psychometric properties. Adolescent and caregiver will complete this measure.
Change from pre therapy to post therapy treatment in adolescent behavior problems as measured by The Achenbach System of Empirically Based Assessments Brief Problem Monitoring (BPM) for 6-18 year old Scales | Pre therapy (at baseline) and post therapy at 24 weeks
  The BPM's Internalizing (INT), Attention Problems (ATT), Externalizing (EXT), and Total Problems (TOT) scales comprise items from the Child Behavior Checklist for Ages 6-18, Teacher's Report Form (TRF), and Youth Self- Report (YSR). The items, scales, and norms are based on decades of research and practical experience, as summarized in the BPM Manual. For this study we will use the youth and caregiver reporting versions.
Change in organizational readiness as measured by Training and Implementation Associates (TIA) Organizational Readiness Measure, Director Form | Pre(baseline) and post organizational consultation (2 weeks)
  This assessment is intended to help TIA identify attitudes, processes and issues that can impact the success of adoption, implementation, and sustainment of a new practice. The information guides our consultation with the agency leaders as we embark on training and implementation of a new evidence-based treatment. The measure focuses on attitudes, knowledge, and current processes, values, and conditions within the agency and workforce.
Dates of the training process as measured by The Training Process Log | 6 months
  The Training Process Log will capture the date that a trainee was hired, the date that the trainee received training, and how the agency handled the period between hiring and the formal training on the evidence-based treatment.
Optimization of technology platform will be measured using the Technology Optimization Log | 4 months
  The Optimization Log will document the additional paths, learning competencies, new simulations, etc., that are created to ensure that all competencies have multiple paths and options for learning.
Competency in evidenced based treatment as measured by CIFFTA Competencies Rating | Pre-training phase and post-training phase (4 weeks later)
  This measure is a modification of the Basic Skills Evaluation Device that was designed to evaluate family therapy competencies and document change. Standard case vignettes are used to elicit interventions that are then rated. The standardization of the clinical situation reduces variability and noise in rating competencies. Our system is tailored to the specific competencies emphasized by CIFFTA but several are core family competencies. These include reframing, blocking negative/hostile interactions, and highlighting caring and protective actions in the family as well as motivational enhancement and engagement interventions.

SECONDARY OUTCOMES:
Therapeutic alliance as measured by the Working Alliance Inventory (WAI) short form | At 5-6 weeks of treatment
  This alliance measure is one of the most recognized and used self-report measures of therapeutic alliance. WAI is a 10-item measure of the quality and strength of the alliance between therapist and client on three dimensions: Goal, Task, and Bond. Adolescents and caregiver will complete this self-report measure.
Satisfaction with the CIFFTA evidenced based treatment as measured by a 10 question survey about satisfaction. | At 5-6 weeks of treatment
  Clients will be asked 10 questions about their satisfaction with the different components of treatment, the involvement of family members, and the inclusion of cultural content in sessions. The degree to which the work was useful will be scored on a 1-5 scale. Adolescent and caregiver will complete it.
Activities related to agency readiness as measured by The Organizational Readiness Consultation Activity Log | Through study completion, an average of 1 year
  The Log will systematically document every activity related to agency readiness and issues that emerge related to agency readiness consultations.
Usefulness of the platform for therapists as measured by Trainee Rating of Usefulness of the Platform and Confidence in Implementing Techniques | At 4 weeks
  The Trainee Rating of Usefulness of the Platform and Confidence in Implementing Techniques is an online measure that is completed after each of the six CIFFTA competencies in the FTTIP online condition. In addition to overall rating of satisfaction, four specific questions will be asked across all modules: How confident are you in your skills at performing the following? How much more training and coaching would you like to receive in this area to master it? How useful was the learning platform in introducing the concepts? How useful was the platform in helping you practice? The responses are rated on a 1-5 scale (e.g., 5 = Very Useful). The responses to these questions were very valuable in the evaluation of the training modules.

CONTACTS AND LOCATIONS:
Overall Officials: David Santisteban, PhD, Principal Investigator — Training and Implementation Associates; Daniel Santisteban, PhD, Study Director — Training and Implementation Associates
Locations (2):
- United States (2):
  - Pacific Clinics, Los Angeles, California
  - Miami Dade County Public Schools, Miami, Florida

IPD SHARING:
Plan to Share IPD: No